CLINICAL TRIAL: NCT04362930
Title: Cohort of Patients With Covid-19 Presenting Neurological or Psychiatric Disorders: An Observational Study of the Covid-19 Neurological and Psychiatric Manifestations
Brief Title: Cohort of Patients With Covid-19 Presenting Neurological or Psychiatric Disorders (CoCo-Neurosciences)
Acronym: CoCo-Neuro
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP200525
Record Dates: First submitted 2020-04-24; First posted 2020-04-27 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-02

CONDITIONS: Neurologic Manifestations; Psychiatric Disorders; COVID-19
Keywords: COVID-19; ENCEPHALOPATHY; ENCEPHALITIS; STROKE; CONFUSION; DELIRIUM; DEPRESSION; POST TRAUMATIC STRESS DISORDER
MeSH Terms: conditions — Neurologic Manifestations; Mental Disorders; COVID-19; Brain Diseases; Encephalitis; Stroke; Confusion; Delirium; Depression; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Neurological and psychiatric impact of COVID-19: Covid-19 impact in neurological or psychiatric manifestations in patients with Covid-19 infection
- Impact of Covid-19 in patients with neurological pathology: patients initially followed for a neurological or psychiatric pathology, suffering from a Covid-19 infection

SUMMARY:
Covid-19 pandemic now affects more than two million people worldwide. The neurotropism of the virus is assumed by its frequent association with neurological symptoms (anosmia, ageusia, headaches) but the extent of the central or peripheral nervous system involvement and the associated symptomatology remain poorly known for now. The main objective of this study is to describe the neurological and psychiatric manifestations occurring in the context of Covid-19 infection in patients hospitalized or followed-up in the APHP.SU hospital group. A better understanding of the neuropsychiatric impairment related to Covid-19 would improve the management of these patients in the acute phase, and knowledge of subsequent complications would allow adapting their rehabilitation and follow-up. The precise phenomenological description of these manifestations and the imaging, biology and neuropathology data will be compiled from the data collected by the physicians in charge of these patients as part of their inpatient or outpatient care. This study will also allow collecting unusual clinical manifestations from patients followed for neurological or psychiatric pathology in hospital departments and presenting a Covid-19 infection, in order to optimize the reorganization of their management, follow-up and rehabilitation in the epidemic context.

DETAILED DESCRIPTION:
Pandemic context In December 2019, the first cases of SARS-CoV-2 coronavirus infection (Covid-19) appeared in Wuhan, Hubei Province, China. The virus quickly spread to other Chinese provinces and then to the rest of the world. The first cases in France were diagnosed on 23 January 2020 in patients who had been in China, and the number of cases rapidly increased to 100 confirmed cases on 29 February 2020. As of 16 April, 106,206 patients had been confirmed, 6,457 patients were hospitalized in intensive care units, and the number of deaths linked to Covid-19 in hospital was 10,643 (government.fr). At the same date, more than 2,065,906 cases were confirmed worldwide, with more than 137,124 deaths (jhu.edu). The most commonly reported clinical manifestation of SARS-CoV-2 infection is an infectious syndrome associated with respiratory signs.

Neurological and psychiatric manifestations of Covid-19 To date, little is known about neurological and psychiatric manifestations of Covid-19. Some authors suggested a significant proportion of patients with central neurological manifestations such as headache, confusion, seizures or strokes. Some cases of COVID-19 encephalitis have also been reported: a case of acute haemorrhagic encephalitis, and a case of encephalitis with seizure and positive SARS-CoV-2 PCR in the CSF. Neurological impairment of Covid-19 has been proposed as a contributing mechanism to respiratory failure in some patients with severe disease. Anosmia and ageusia are now recognized as common symptoms of the infection. Cases of Guillain-Barré syndrome and probable myelitis (without radiological confirmation) have also been described. Myalgia is frequently reported in patients with Covid-19 infection, but no cases of documented myopathy have been reported to date.

Patients with Covid-19 infection may also present systemic encephalopathy in the context of severe respiratory failure, associated organ failure (renal, hepatic), and iatrogenicity.

Patients hospitalized in intensive care unit for severe forms of the infection frequently present with confusion, and sometimes persistent cognitive disorders such as a dysexecutive syndrome, attention disorders, spatio-temporal disorientation. A high frequency of clinical signs of cortico-spinal bundle damage and leptomeningeal contrast images on cerebral MRI has also been reported.

Regarding psychiatric manifestations, a high prevalence of anxiety disorders and depressive syndromes was noted in patients with Covid-19. Post-traumatic stress disorder may also occur in these patients, particularly those who have suffered from severe forms of stress and have been hospitalized in intensive care units.

SARS-CoV-2 is a member of the coronavirus family and bears a strong similarity to other coronaviruses such as SARS-CoV or MERS-CoV. Clinical and preclinical knowledge of other coronaviruses suggests neurotropism of viruses of this family. In particular, infection with SARS-CoV-2 or NCoV-OC43 may cause encephalitis or encephalomyelitis. The SARS-CoV-2 virus adheres to cell membranes by interaction with ACE2 receptors, which are highly expressed on the surfaces of neurons and glial cells. The ACE2 receptor is particularly expressed in the brainstem and in regions involved in cardiovascular control including the paraventricular nucleus, the nucleus of the solitary tract. The virus could reach the nervous system via systemic circulation (viremia) or via ethmoidal microcirculation via the olfactory epithelium. Indeed, animal studies have shown that SARS-Cov can invade the brain via the olfactory epithelium via the nasal route and cause neuronal death. The virus could also infect the brain through trans-synaptic transmission from the olfactory epithelium through the ethmoidal floor to the olfactory bulb. Another mechanism of neurological damage related to Covid-19 infection could be the initiation of an immune reaction with the release of cytokines and other inflammatory proteins, leading to a breakdown of the blood-brain barrier, which amplifies neuro-inflammatory processes. Systemic inflammation and cytokines may also promote ischemic stroke. Severe coagulopathies have been reported.

Covid-19 and pre-existing neurological and psychiatric disorders SARS-CoV-2 infection could lead to the aggravation of certain pre-existing neurological and psychiatric disorders, but the potential impact of the infection in the short, medium and long term on these pathologies is still unknown.

Indeed, infections are a classic aggravating factor in many neurological pathologies, such as autoimmune pathologies, metabolic pathologies, and also neurodegenerative pathologies. Brain inflammation is recognised as an important mechanism of neurodegenerative pathologies and has also been implicated in psychiatric pathologies such as schizophrenia and depression.

Patients with cardiac or respiratory damage, particularly in the context of neuro-muscular pathologies, could particularly develop severe forms of infection. Patients with neurodegenerative pathologies often represent an elderly population, and therefore also at risk of severe forms of infection. Patients followed for inflammatory or neuro-oncological pathologies and undergoing immunosuppressive treatments or chemotherapy also represent a at-risk population. SARS-CoV-2 infection could also worsen certain psychiatric pathologies.

Public interest research Neurological and psychiatric manifestations have been reported in patients with Covid-19 but the different neuropsychiatric expressions of Covid-19 infections are currently not well characterized.

A better understanding of the neurological and psychiatric impairment related to Covid-19 could improve management of the patients in the acute phase.

Knowledge of neurological and psychiatric complications subsequently occurring would allow adapting the follow-up of these patients. The inclusion of prospective long-term follow-up data is crucial in the overall understanding of the neuropsychiatric disorders of Covid-19. Neurological complications are likely to occur at a distance from the infection or to be lately diagnosed, for instance, in patients who have been in intensive care. The collection of data from the rehabilitation follow-up of these patients is crucial in this context.

The precise phenomenological description of these manifestations and the collection of imaging, biological and neuropathological data may also allow establishing hypotheses on the pathophysiology of the neurological damage caused by Covid-19.

The impact of Covid-19 infection on pre-existing neurological and psychiatric pathologies is not known. This knowledge would optimize the reorganization of the management, follow-up and rehabilitation of these patients in the epidemic context.

In this observational, retrospective, multicentre study, the investigators aim at i) describing the clinical and paraclinical manifestations of patients with neurological or psychiatric manifestations of Covid-19 infection, and ii) describing changes in the clinical trajectories of patients with Covid-19 infection, initially followed for neurological or psychiatric pathologies.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 years or over
* Patient followed for a neurological or psychiatric pathology OR Patient consulting and presenting a neurological or psychiatric impairment AND
* Presenting a COVID-19 infection defined by at least one of the following three criteria:

  * Biological diagnosis by any method for direct detection of the virus (Covid-19 positive PCR) or recent infection (serology)
  * Typical chest imaging (CT scan or X-ray) in an epidemic area
  * Clinical-biological data leading to a strong suspicion of current or past Covid-19 infection
* Non-opposition of the participant, relative or guardian to the research

Exclusion Criteria:

* Patient under safety measure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Covid-19 infection showing neurological or psychiatric symptoms and patients initially followed for a neurological or psychiatric pathology, suffering from a Covid-19 infection
Sampling Method: Non-Probability Sample
Enrollment: 730 (Actual)
Dates: Start 2020-04-27 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Central or peripheral neurological symptoms or psychiatric symptoms observed in patients with Covid-19 | 12 months
  Frequency of central or peripheral neurological or psychiatric symptoms observed in patients with COVID-19

SECONDARY OUTCOMES:
Progression of pre-existing neurological or psychiatric pathologies | 12 months
  Impact on neurological or psychiatric disease trajectories assessed by severity scores or subjective progression (improved, stable, impaired) during and after COVID-19 pathology in patients with pre-existing neurological and psychiatric diseases

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Pitié Salpétrière, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pitron V, Cantenys W, Herbelin A, Bottemanne H, Dzierzynski N, Caumes E, Mathian A, Amoura Z, Allenbach Y, Cacoub P, Parrot A, Rotge JY, Fossati P. Factors Associated With Posttraumatic Stress Symptoms 3 and 6 Months After Hospitalization for COVID-19: A Longitudinal Multicenter Study. J Clin Psychiatry. 2022 Dec 7;84(1):21m14277. doi: 10.4088/JCP.21m14277. PMID 36479951
- See also: CoCo-Neurosciences project is described on the Paris Brain Institute website — https://icm-institute.org/